CLINICAL TRIAL: NCT00167973
Title: A Prospective Registry of European Hemophilia B Patients Receiving BeneFIX®(Nonacog Alfa, Recombinant Human Factor IX) for Usual Use
Brief Title: Prospective Registry of European Hemophilia B Patients Receiving BeneFIX® for Usual Use
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3090A-101039
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Hemophilia B
Keywords: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is an open-label multi-center Registry in patients with hemophilia B receiving BeneFIX. All patients who begin treatment with BeneFIX in European Union countries, will be eligible for participation. Patient demographics will be collected at baseline for all patients. A baseline FIX activity and Bethesda assay for inhibitor based on historical data should be recorded if available. Adverse events as defined in the protocol will also be reported on the appropriate forms. Data will be collected from patients on an ongoing basis to ensure that information is being captured for each patient being treated with BeneFIX.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hemophilia B scheduled to begin treatment with BeneFIX are eligible for Registry enrollment

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All EU patients beginning treatment with BeneFIX
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2002-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Observation for safety | Study Duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial mANAGER, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Sweden, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com
Locations (83):
- Vienna, Austria
- Belgium (4):
  - Brussels
  - Edegem
  - Leuven
  - Montegnée
- France (21):
  - Amiens
  - Angers
  - Caen
  - Chambéry
  - Grenoble
  - Le Chesnay
  - Le Kremlin-Bicêtre
  - Liffré
  - Limoges
  - Lyon
  - Marseille
  - Montmorency
  - Montpellier
  - Nantes
  - Nevers
  - Nice
  - Osséja
  - Paris
  - Rouen
  - Saint-Priest-en-Jarez
  - Tours
- Germany (3):
  - Erlangen, Bavaria
  - Hamburg, Hamburg
  - Münster, North Rhine-Westphalia
- Italy (16):
  - Ancona, AN
  - Bari, BA
  - Catania, CT
  - Catanzaro, CZ
  - Milan, MI
  - Palermo, PA
  - Pescara, PE
  - Parma, PR
  - Reggio Calabria, RC
  - Sassari, SS
  - Napoli
  - Padua
  - Palermo
  - Perugia
  - Roma
  - Vicenza
- Netherlands (6):
  - Amsterdam
  - Breda
  - Eindhoven
  - Maastricht
  - Nijmegen
  - Utrecht
- Coimbra, Portugal
- Spain (13):
  - Almería
  - Barcelona
  - Burgos
  - Cadiz
  - Esplugues de Llobregat
  - Madrid
  - Mérida-Badajoz
  - Santander
  - Seville
  - Valencia
  - Valladolid
  - Vitoria-Gasteiz
  - Zaragoza
- Sweden (2):
  - Malmo
  - Stockholm
- United Kingdom (16):
  - Truro, Cnwll
  - London, Gt Lon
  - Manchester, Gt Man
  - Edinburgh, Loth
  - Liverpool, Mersyd
  - Sheffield, Mersyd
  - Oxford, Oxon
  - Sheffield, Syorks
  - Cardiff, W Glam
  - Birmingham, Wstmid
  - Wolverhampton, Wstmid
  - Leeds, Wyorks
  - London
  - Plymouth
  - Poole
  - Sheffield

REFERENCES:
- [Derived] Rendo P, Smith L, Lee HY, Shafer F. Nonacog alfa: an analysis of safety data from six prospective clinical studies in different patient populations with haemophilia B treated with different therapeutic modalities. Blood Coagul Fibrinolysis. 2015 Dec;26(8):912-8. doi: 10.1097/MBC.0000000000000359. PMID 26196195